CLINICAL TRIAL: NCT05754489
Title: Exercise Oxygen Kinetic and Cardiac Output in Hypertrophic Cardiomyopathy: a Multicenter Prospective Cardiopulmonary Exercise Testing Study
Brief Title: Exercise Oxygen Kinetic and Cardiac Output in Hypertrophic Cardiomyopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Azienda Sanitaria Universitaria Giuliano Isontina [ASUGI], Università di Trieste, Italy (Unknown); Azienda Ospedaliera "Sant'Andrea" (Other)
Responsible Party: Sponsor
Other Study IDs: CCM 1750
Record Dates: First submitted 2023-02-15; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Cardiopulmonary Exercise Test; Hypertrophic Cardiomyopathy; Cardiac Output Measurement
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fatigue and dyspnea that reduce exercise performance are common symptoms in patients with hypertrophic cardiomyopathy. Since the cause of this functional limitation has not yet been described, this study aims to evaluate the cardiopulmonary parameters measured at cardiopulmonary exercise test in combination with those obtained by non-invasive measurement of cardiac output by impedance (Physioflow) and echocardiography. These results will help to better define the mechanisms underlying limitation in these patients, also in relation to the degree of LVOT obstruction.

The aim of the present study is to assess the cardiopulmonary response to exercise in patients with hypertrophic cardiomyopathy, based on the degree of LVOT obstruction, by adding non-invasive measurement of cardiac output by Physioflow and echocardiographic parameters to the cardiopulmonary exercise test parameters associated with stroke volume and cardiac output (ie. VO2/WR, O2pulse) Consecutive patients with a previous diagnosis of hypertrophic cardiomyopathy on optimised medical therapy will be enrolled to perform a cardiopulmonary exercise test with simultaneous measurement of cardiac output and an exercise echocardiogram for clinical routine.

ELIGIBILITY:
Inclusion Criteria:

* hypertrophic cardiomyopathy diagnosis

Exclusion Criteria:

* use of long-term oxygen therapy;
* presence of comorbidities affecting the ability to perform cardiopulmonary exercise test or interfering with exercise performance;
* concomitant at least moderate chronic obstructive pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with a previous diagnosis of hypertrophic cardiomyopathy in optimised medical therapy will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
cardiac output measurement | immediately after the evaluation
  Evaluate cardiopulmonary exercise test parameters associated with stroke volume and cardiac output (ie. VO2/WR, O2pulse) with the addition of non-invasive measurement of cardiac output using Physioflow.

SECONDARY OUTCOMES:
Correlation with echocardiographic variables | immediately after the evaluation
  Correlate functional and metabolic data with echocardiographic variables collected at rest and under stress.

CONTACTS AND LOCATIONS:
Overall Officials: Piergiuseppe Agostoni, Prof., Principal Investigator — Centro Cardiologico Monzino
Locations (3):
- Italy (3):
  - Centro Cardiologico Monzino, Irccs, Milan
  - Azienda Ospedaliera Sant'Andrea, Rome
  - Azienda Sanitaria Universitaria Giuliano Isontina [ASUGI], Trieste

IPD SHARING:
Plan to Share IPD: Undecided